CLINICAL TRIAL: NCT05006274
Title: Evaluation of Intraoperative Soft-tissue Balance and Postoperative Functional Recovery After Total Knee Arthroplasty
Brief Title: Intraoperative Soft Tissue Balance in TKA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington Hospital Healthcare System (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Alexander Sah, MD, Physician and Research Chair, Institute for Joint Restoration and Research, Washington Hospital Healthcare System
Other Study IDs: IRU2018-51K
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group 1-Traditional soft tissue balance: Patients in group 1 will receive traditional, manual soft-tissue balancing during surgery. For the purpose of the study, the balance will be quantitatively assessed at the end of the case, by means of surgeon-blinded VERASENSE measurements before and after cementation.
  Interventions: Device: Persona Trabecular Metal Tibia; Device: Verasense technology; Device: MUVR
- Group 2-Soft tissue balance using VERASENSE: For the patients in Group 2, intra-operative sensor feedback will be used in creating a quantitatively balanced knee (VERASENSE, OrthoSensor Inc.). Thereby, a quantitatively balanced knee is characterized by a mediolateral load differential below 15lbs at 10-45-90 degrees of flexion.
  Interventions: Device: Persona Trabecular Metal Tibia; Device: Verasense technology; Device: MUVR

INTERVENTIONS:
Device: Persona Trabecular Metal Tibia — Total knee arthroplasty
Device: Verasense technology — Instrumented tibial trial component
Device: MUVR — Knee motion and gait sensing wearable device

SUMMARY:
The purpose of this evaluation is to evaluate the intraoperative soft tissue balance as assessed by the Orthosensor device, to measure the perioperative gait and function with the Muvr tracking device, and to correlate this soft tissue balance with early functional outcomes in the Persona total knee system.

DETAILED DESCRIPTION:
This is a single surgeon, prospective, controlled study consisting of 50 patients with a primary indication of OA who are eligible for primary total knee arthroplasty using the Persona total knee system.

The patients are equally divided in two groups; patients in group 1 will receive traditional, manual soft-tissue balancing during surgery. For the purpose of the study, the balance will be quantitatively assessed at the end of the case, by means of surgeon-blinded VERASENSE measurements before and after cementation. For the patients in Group 2, intra-operative sensor feedback will be used in creating a quantitatively balanced knee (VERASENSE, OrthoSensor Inc.). Thereby, a quantitatively balanced knee is characterized by a mediolateral load differential below 15lbs at 10-45-90 degrees of flexion.

Post-operatively, the patients will be evaluated using the Muvr device at the day of surgery, day of discharge and 2, 6, and 12 weeks, and 1 year postoperatively. This device will provide quantitative feedback on different gait metrics as well as function during activities of daily living such as stair climbing / stair descent, walking, and timed get up and go testing.

During each post-operative visit, the following metrics will be recorded:

* Active and passive range of motion
* Implant alignment
* Patient reported outcomes by means of Knee Society Score (KSS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Forgotten Joint Score (FJS)

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a primary indication of osteoarthritis and is eligible for primary total knee arthroplasty using the Persona total knee system
2. Patient is willing and able to provide written Informed Consent prior to study surgery
3. Patient is willing and able to complete scheduled study procedures and follow-up evaluations as described in the Informed Consent Form

Exclusion Criteria:

1. Patient does not have a primary indication of osteoarthritis
2. Patient does not have access to internet or mobile device or understand how to use phone/app
3. Patient is not eligible or will not receive the Persona total knee system
4. Patient has not provided written Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy individuals having elective primary knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Active and passive range of motion | 2 weeks
  Flexion and extension measurements of knee
Active and passive range of motion | 6 weeks
  Flexion and extension measurements of knee
Active and passive range of motion | 12 weeks
  Flexion and extension measurements of knee
Active and passive range of motion | 1 year
  Flexion and extension measurements of knee
Implant alignment | 2 weeks post-operatively
  Radiographic assessments
Implant alignment | 6 weeks post-operatively
  Radiographic assessments
Implant alignment | 12 weeks post-operatively
  Radiographic assessments
Implant alignment | 1 year post-operatively
  Radiographic assessments
Knee Society Score (KSS) | 2 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-100, higher score better.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 2 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-96, lower score means less disability
Forgotten Joint Score (FJS) | 2 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-100, 100 being better score
Knee Society Score (KSS) | 12 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-100, higher score better.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-96, lower score means less disability
Forgotten Joint Score (FJS) | 12 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-100, 100 being better score
Knee Society Score (KSS) | 52 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-100, higher score better.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 52 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-96, lower score means less disability
Forgotten Joint Score (FJS) | 52 weeks post-operatively
  Patient-reported outcome surveys assessing pain and function after total knee arthroplasty. Range 0-100, 100 being better score

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: No